CLINICAL TRIAL: NCT02728219
Title: A Prospective Randomized Trial Comparing Treatment of Recurrent HCC With Repeat Hepatectomy,and Transcatheter Arterial Chemoembolization (TACE) With AFP Conversion
Brief Title: Comparison of Treatment of Recurrent HCC With Repeat Hepatectomy,and TACE With AFP Conversion
Acronym: HCCTACEAFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012ZX10002016007002
Record Dates: First submitted 2016-03-28; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Recurrent Hepatocellular Carcinoma
Keywords: Recurrent Hepatocellular Carcinoma; transcatheter arterial chemoembolization; AFP conversion
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hepatectomy (Experimental): Comparison of Treatment of recurrent hepatocellular carcinoma with repeat hepatectomy,and transcatheter arterial chemoembolization (TACE) with AFP conversion
  Interventions: Procedure: TACE
- TACE (Active Comparator)
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: TACE — In this study we prospectively select some early diagnosed recurrent HCC patients after radical resection with AFP conversion, then they will be treated with transcatheter arterial chemoembolization (TACE)
  Other Names: transcatheter arterial chemoembolization
  Arms: hepatectomy
Procedure: Hepatectomy — Repeat Hepatectomy after postoperation recurrence
  Arms: TACE

SUMMARY:
The purpose of this study is to compare the treatment of recurrent hepatocellular carcinoma with repeat hepatectomy,and transcatheter arterial chemoembolization (TACE) with AFP conversion.

DETAILED DESCRIPTION:
Though many HCC patients have been benefited from hepatectomy treatment, still the high recurrence rate after the hepatectomy led to limited effectiveness.

This is the first study in same case system on comparison of effectiveness among repeat hepatectomy, and TACE with AFP conversion.

ELIGIBILITY:
Inclusion Criteria:

1. via clinical diagnosis and confirm it is early recurrent liver cancer with AFP conversion, and not accept any anticancer treatment.
2. age:18-70years
3. better liver function (Child-Pugh，class A or B)

Exclusion Criteria:

1. reject to attend；
2. impossible to come to our hospital for physical examination regularly.
3. cancer epitome、seed focus、lymph node or distant metastasis
4. Blood clotting function hindrance;
5. serious heart、lung、kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China